CLINICAL TRIAL: NCT04350411
Title: Comparison of PEAK PlasmaBlade™ to Conventional Diathermy in Abdominal Based Free Flap Breast Reconstruction - a Single Centre, Double Blinded Randomised Controlled Trial
Brief Title: Comparison of PEAK PlasmaBlade™ to Conventional Diathermy in Abdominal Based Free Flap Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Collaborators: Mid Essex Hospital NHS Trust (Other); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 16/17 086
Record Dates: First submitted 2020-04-06; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Breast Reconstruction; Breast Cancer
Keywords: Electrosurgery; Conventional diathermy; PEAK PlasmaBlade™; Deep Inferior Epigastric Perforator (DIEP) flap; Drain; Seroma
MeSH Terms: conditions — Breast Neoplasms; Hyperthermia; Seroma

STUDY DESIGN:
Intervention Model Description: Patients randomised between having their procedure performed with one of two different electrosurgery devices
Who Masked: Participant, Investigator
Masking Description: Patients and investigator collecting data were both blinded for which machine was used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional diathermy (Experimental): DIEP/ MS-TRAM breast reconstruction free flap raise performed with conventional diathermy
  Interventions: Device: Conventional diathermy
- PEAK PlasmaBlade™ (Experimental): DIEP/ MS-TRAM breast reconstruction free flap raise performed with PEAK PlasmaBlade™
  Interventions: Device: PEAK PlasmaBlade™

INTERVENTIONS:
Device: Conventional diathermy — Abdominal free flap raise performed with conventional diathermy. Settings: cutting 40 Watt, coagulation 40 Watt.
  Arms: Conventional diathermy
Device: PEAK PlasmaBlade™ — Abdominal free flap raise performed with PEAK PlasmaBlade™ Settings: cutting 7 (35 Watt), coagulation 7 (35 Watt)
  Arms: PEAK PlasmaBlade™

SUMMARY:
Electrosurgery allows for dissection with simultaneous haemostasis. One of its disadvantages is that the heat production can cause injury to the surrounding tissue which may result in wound healing problems and an increased rate of seromas.

The PEAK PlasmaBlade™ (PPB) is a new electrosurgery device which may overcome this by having the ability to operate on a lower temperature, therefore reducing collateral thermal damage.

Different experimental studies in both animal and human models comparing the PEAK PlasmaBlade™ and other surgical dissection devices for incisions have shown a reduction in width of zone of thermal injury, reduction in wound inflammation, increased wound strength and reduced scaring in favour of the PEAK PlasmaBlade™ and comparable to scalpel incisions. A prospective clinical study published by Dogan et al. in 2013, including 46 consecutive breast cancer patients receiving a modified radical mastectomy either with the conventional diathermy (n=22) or the PEAK PlasmaBlade™ (n=24), showed a statistically significant reduction in wound fluid production (p=0.025), leading to earlier drain removal (p=0.020) in the PEAK PlasmaBlade™ group.

Comparable to oncological breast surgery, prolonged drain requirements for high wound fluid production and seromas are often experienced in the abdominal donor side after deep inferior epigastric perforator/ muscle sparing transverse rectus abdominis muscle flap (DIEP/MS-TRAM) breast reconstruction. To evaluate the effects of the PEAK PlasmaBlade™ for abdominal dissection in autologous breast reconstruction on wound fluid production and complications such a seroma, this double blinded randomised controlled clinical trial was conducted.

It was hypothesised the use of the PEAK PlasmaBlade™ for the harvest of the DIEP/ MS-TRAM flap would result in 1) a shorter abdominal drains requirement (days); 2) a lower total drainage volume (mL) from the abdominal drains; 3) lower levels of inflammatory cytokines in the drain fluid and 4) less and smaller seromas would be identified using ultrasound in the follow-up period.

DETAILED DESCRIPTION:
The study was conducted between November 2016 and May 2018 in a single centre, St. Andrew's Centre for Plastic Surgery and Burns in Broomfield Hospital, in Chelmsford United Kingdom, including all immediate and delayed DIEP/MS-TRAM patients of two senior plastic surgeons, who agreed to participate and met the in-/exclusion criteria. All participants signed an informed consent. Randomisation was performed using the Trans European Network for Clinical Trials Service (TENALEA), which is an internet-based randomisation system. Patients were either allocated to the 'Group A - diathermy' or 'Group B - PEAK PlasmaBlade™. Blinding was broken after the last patient had completed the 6-week follow-up period.

All patients underwent a standardised DIEP or MS-TRAM breast reconstruction procedure. A scalpel was used to make the skin incision to the depth of the dermis. The raising of the flap was subsequently done either using the PEAK Plasma Blade™ or conventional diathermy. Before the abdominal closure two 15 French Blake drains were inserted and secured to the skin with a 2.0 Silk suture and connected to a low vacuum wound drainage system (85 kPa/neg 100mmHg). Every patient would wear an abdominal binder (9-inch, Marena) for 6 weeks post-operatively. Data on drain requirement, total daily abdominal drainage, pain, mobility and complications were collected during the inpatient stay. On day 0,1 and 2 also abdominal drain fluid was obtained. This was stored in labelled 1.5mL Eppendorf tubes in a -80°C freezer. The samples were sent to Myriad RBM, Inc. a clinical laboratory improvement amendments (CLIA) certified biomarker testing laboratory located in Austin, Texas (United States) for inflammatory cytokine analysis. Abdominal drains were removed when draining 30mL or less in 24 hours. Following discharge, patients were seen in the outpatient department after two and six weeks. At both follow-up appointments, data on complications were recorded. Also an abdominal ultrasound was performed using the V-Universal™ Stand portable ultrasound machine (SonoSite, Inc) to identify and measure abdominal seroma collections. Seromas were only aspirated if they were causing discomfort to the patient. After completion of the 6-week follow-up period patients were discharged from the study. All data were collected by the blinded principle study investigator and logged onto an electronic database.

Data from an in the investigator's unit conducted pilot study on drain requirement was used to perform a power calculation.This results in a minimal sample size of 53 patients for each group (106 overall).

Normal distribution was evaluated using the Shapiro-Wilk test, following this continuous data was analysed using the independent sample t-test or Mann-Whitney U Test to identify a statistically significant difference between the two groups. All right skewed was log transformed, if this resulted in a normal distribution the independent samples t-test was used to determine statistical significance. For categorical data the Pearson Chi-Square Test for numbers over 5 was used. If the count was equal to or less than 5 the Fisher's Exact Test was used to determine statistical significance. A value below or equal to 0.05 (2-tailed) was considered to be statistically significant. Linear regression (Cox proportional hazard model) was used to identify significant determinants for the time to drain removal. Variables that had a significant p-value in the univariate analysis were included in a multivariable analysis. Significant determinants could indicate confounding factors for which would be corrected. Logistic regression was used to identify determinants for complications and the presence of seroma at the 2- and 6-week abdominal ultrasound scan. Variables that had a significant p-value in the univariate analysis were included in multivariable analysis, if none of the determinates were significant p values <0.10 were included in the multivariable analysis. Significant determinants could indicate confounding factors for which would be corrected.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18-80 years, able to consent
* Unilateral immediate or delayed DIEP/ MS-TRAM breast reconstruction
* BMI >20

Exclusion Criteria:

* Children (<18 years) and adults older than 80 years
* Bilateral or bi-pedicled DIEP/MS-TRAM breast reconstruction
* BMI <20
* Diabetic
* Immune-suppression
* Clotting disorders
* On steroid medication
* Pregnancy
* Active smoking

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females undergoing immediate or delayed abdominal based free flap breast reconstruction
Enrollment: 108 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Number of days the abdominal drains were required | Drain requirement from the day of operation (day 0) until the day the drain was removed when producing 30ml or less/ 24 hours
  Number of days post operative

SECONDARY OUTCOMES:
Flap raise time | Data recorded during operation
  Time required to raise abdominal flap (minutes)
Weight of abdominal flap | Data recorded during operation
  Weight of raised abdominal flap in grams
Inflammatory markers in abdominal drain fluid on day 0,1 and 2 | Drain fluid on day 0, 1 and 2
  Inflammatory markers in abdominal drain fluid: TNF-alpha, IL-4, IL-6,IL-8, IL-10, IL-18, MIP-1 alpha, MIP-1 beta, MCP-1
Pain score | Recorded twice a day (morning and afternoon) while an inpatient (between 3 - 14 days)
  Numerical rating scale (NRS) 0 to 10 (with 0 being no pain and 10 the worse pain imaginable)
Mobility | While an inpatient (between 3 - 14 days)
  Number of steps a day
Total abdominal drain fluid output | Total amount of abdominal drain fluid collected at time of drain removal (between 3 - 14 days post-operatively)
  Total amount of fluid drained from abdominal wound (millilitres) during admission
Complications | In the 6-week follow-up period
  Number of complications during the study experienced by each patient (for example: Flap problems, haematoma, delayed abdominal wound healing, seroma)
Interventions for complications | In the 6-week follow-up period
  Number of interventions required to deal with complication for each patient (for example needle aspiration, surgery, iv antibiotics)
Seroma presence on abdominal ultrasound | At the 2- and 6-week follow-up appointments
  Abdominal ultrasound to identify
Size of seroma collection on abdominal ultrasound | At the 2- and 6-week follow-up appointments
  Size (length, width and depth was measured and used to estimate the size using the formula of half an ellipse)

CONTACTS AND LOCATIONS:
Overall Officials: Thessa R Friebel, MSc, Principal Investigator — Mid Essex NHS trust; Matthew Griffiths, MBBS, MD, Study Director — Mid Essex NHS trust; Selim Cellek, MD, PhD, Study Director — Anglia Ruskin University
Locations (1):
- Mid Essex NHS trust, Chelmsford, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the IPD

REFERENCES:
- [Background] Massarweh NN, Cosgriff N, Slakey DP. Electrosurgery: history, principles, and current and future uses. J Am Coll Surg. 2006 Mar;202(3):520-30. doi: 10.1016/j.jamcollsurg.2005.11.017. No abstract available. PMID 16500257
- [Background] Yilmaz KB, Dogan L, Nalbant H, Akinci M, Karaman N, Ozaslan C, Kulacoglu H. Comparing scalpel, electrocautery and ultrasonic dissector effects: the impact on wound complications and pro-inflammatory cytokine levels in wound fluid from mastectomy patients. J Breast Cancer. 2011 Mar;14(1):58-63. doi: 10.4048/jbc.2011.14.1.58. Epub 2011 Mar 31. PMID 21847396
- [Background] Loh SA, Carlson GA, Chang EI, Huang E, Palanker D, Gurtner GC. Comparative healing of surgical incisions created by the PEAK PlasmaBlade, conventional electrosurgery, and a scalpel. Plast Reconstr Surg. 2009 Dec;124(6):1849-1859. doi: 10.1097/PRS.0b013e3181bcee87. PMID 19952641
- [Background] Ruidiaz ME, Messmer D, Atmodjo DY, Vose JG, Huang EJ, Kummel AC, Rosenberg HL, Gurtner GC. Comparative healing of human cutaneous surgical incisions created by the PEAK PlasmaBlade, conventional electrosurgery, and a standard scalpel. Plast Reconstr Surg. 2011 Jul;128(1):104-111. doi: 10.1097/PRS.0b013e31821741ed. PMID 21701326
- [Background] Dogan L, Gulcelik MA, Yuksel M, Uyar O, Erdogan O, Reis E. The effect of plasmakinetic cautery on wound healing and complications in mastectomy. J Breast Cancer. 2013 Jun;16(2):198-201. doi: 10.4048/jbc.2013.16.2.198. Epub 2013 Jun 28. PMID 23843853